CLINICAL TRIAL: NCT06185699
Title: Could Wearing Face Mask During the Pandemic Have Created An Environment for Demodex Mites?
Brief Title: Could Wearing Face Mask Have Affected Demodex Parasite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurhan Döner Aktaş (Other)
Responsible Party: Sponsor-Investigator, Nurhan Döner Aktaş, dermatology specialist, principal investigator, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2021-KAE-0023
Record Dates: First submitted 2023-12-01; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Pandemic, COVID-19; Demodex Infestation
Keywords: Covid-19; demodex; mask
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Individuals (ı) who wore N95/FFP2 masks during the whole working hours, and only took off it for less than 1 hour; (ıı) those who wore a 3-ply surgical mask during all working hours, only took it off for less than 1 hour and (ııı) people who wore a 3-ply surgical mask for less than 3 days a week, less than 2 hours a day and spending time mostly at home during the day or plus those who worked alone all day in their rooms and who wear a 3-ply surgical mask for less than 1 hour during the day as required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- N95/FFP2 masks during the whole working hours, and only took off it for less than 1 hour (Other): Individuals (ı) who wore N95/FFP2 masks during the whole working hours, and only took off it for less than 1 hour. In order to detect the presence of Demodex mites, standard superficial skin biopsy (SSSB) was applied
  Interventions: Diagnostic Test: standard superficial skin biopsy (SSSB)
- 3-ply surgical mask during all working hours, only took it off for less than 1 hour (Other): Individuals who wore a 3-ply surgical mask during all working hours, only took it off for less than 1 hour.In order to detect the presence of Demodex mites, standard superficial skin biopsy (SSSB) was applied
  Interventions: Diagnostic Test: standard superficial skin biopsy (SSSB)
- control (who rarely used masks under pandemic conditions) (Other): people who wore a 3-ply surgical mask for less than 3 days a week, less than 2 hours a day and spending time mostly at home during the day or plus those who worked alone all day in their rooms and who wear a 3-ply surgical mask for less than 1 hour during the day as required. In order to detect the presence of Demodex mites, standard superficial skin biopsy (SSSB) was applied
  Interventions: Diagnostic Test: standard superficial skin biopsy (SSSB)

INTERVENTIONS:
Diagnostic Test: standard superficial skin biopsy (SSSB) — standard superficial skin biopsy (SSSB) was applied to the face that was wiped with dry sterile gauze after dropping cyanoacrylate by marking 1 cm2 area on the slide that was wiped with dry sterile gauze from 3 areas of the face, right cheek, nose and the mid-forehead. After the slide was left for 60 seconds and slowly removed from the face, immersion oil was dripped onto the slide and covered with a coverslip, and Demodex mites were counted first under the light microscope at x10 and then x20 magnification (Demodex foliculorum and brevis were not differentiated). The process was repeated for each region.

SUMMARY:
This study aimed to examine whether wearing masks by healthy individuals during the Covid-19 pandemic created an environment for Demodex mites, by comparing it with the control group. In order to detect the presence of Demodex mites, standard superficial skin biopsy (SSSB) was applied to the face

DETAILED DESCRIPTION:
The study was carried out on March 15.2021 and the data collection was completed within 6 months. For the randomization of the participants, they were first stratified according to age and then the participants were selected according to the simple randomization table and included in the study.The sample of the study was calculated to be at least 48 people for each group, with the power of the test being approximately 80,151%. Ethics committee approval of the study was obtained from the clinical research ethics committee of Katip Çelebi University with no: 27 on 11.03.2021. A total of 144 people who met the inclusion criteria, 48 individuals for each group, were included in the study. The study was conducted in accordance with the principles of the Declaration of Helsinki. Participants were included in the study after signing the informed consent form. The exclusion criteria included having dermatosis (acne, acne rosacea, seborrheic dermatitis) and/or other dermatological diseases associated with the presence of Demodex mites, receiving or having been receiving treatment for Demodex-associated dermatosis (topical and/or systemic), using face wash gel and/or cologne, which prevents the life of Demodex mites, cosmetic cream with pore-clogging feature, applying disinfectant; being obese (BMI> 30), consuming regular alcohol use, and taking oral therapy that suppresses the immune system, or using creams with immunological effects when applied topically on the face as well as developing any skin complaints with wearing masks, Individuals who wore N95/FFP2 masks during the whole working hours, and only took off it for less than 1 hour; (ıı) those who wore a 3-ply surgical mask during all working hours, only took it off for less than 1 hour and (ııı) people who wore a 3-ply surgical mask for less than 3 days a week, less than 2 hours a day and spending time mostly at home during the day or plus those who worked alone all day in their rooms and who wear a 3-ply surgical mask for less than 1 hour during the day as required. The third group represented the control group (the control group was comprised of individuals who presented to the hospital during the study period, since there was no one without mask during the day). Participants were included in the study after signing the informed consent form. The sociodemographic characteristics, including age, gender and occupation; cigarette use, alcohol use, the past medical history, face washing habits (only water, water and soap, non-specific face wash product) and dermatological examination, whether the skin is oily or dry-normal, and Fitzpatrick skin typing were determined. In order to detect the presence of Demodex mites, standard superficial skin biopsy (SSSB) was applied to the face that was wiped with dry sterile gauze after dropping cyanoacrylate by marking 1 cm2 area on the slide that was wiped with dry sterile gauze from 3 areas of the face, right cheek, nose and the mid-forehead. After the slide was left for 60 seconds and slowly removed from the face, immersion oil was dripped onto the slide and covered with a coverslip, and Demodex mites were counted first under the light microscope at x10 and then x20 magnification (Demodex foliculorum and brevis were not differentiated). The process was repeated for each region. The presence of Demodex mites in each region and its number, if any, were written on the inquiry form.

ELIGIBILITY:
Inclusion Criteria:

Individuals (ı) who wore N95/FFP2 masks during the whole working hours, and only took off it for less than 1 hour; (ıı) those who wore a 3-ply surgical mask during all working hours, only took it off for less than 1 hour (ııı) people who wore a 3-ply surgical mask for less than 3 days a week, less than 2 hours a day and spending time mostly at home during the day or plus those who worked alone all day in their rooms and who wear a 3-ply surgical mask for less than 1 hour during the day as required.

(The third group represented the control group (the control group was comprised of individuals who presented to the hospital during the study period, since there was no one without mask during the day).

Exclusion Criteria:

* Having dermatosis (acne, acne rosacea, seborrheic dermatitis) and/or other dermatological diseases associated with the presence of Demodex mites, receiving or having been receiving treatment for Demodex-associated dermatosis (topical and/or systemic)
* Using face wash gel and/or cologne, which prevents the life of Demodex mites, cosmetic cream with pore-clogging feature, applying disinfectant
* Being obese (BMI> 30)
* Consuming regular alcohol use,
* Taking oral therapy that suppresses the immune system, or using creams with immunological effects when applied topically on the face
* Developing any skin complaints with wearing masks.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
presence of demodex mites | 6 month
  The presence of Demodex mites was detected by the standard superficial skin biopsy (SSSB) from 3 regions of the face ( the right cheek, the nose, the mid-forehead).

CONTACTS AND LOCATIONS:
Overall Officials: Nurhan Döner Aktaş, Specialist, Principal Investigator — Izmir Katip Celebi University Atatürk Research and Training Hospital dermatology Department
Locations (1):
- Izmir Katip Çelebi University Atatürk Research and Trainig Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No